CLINICAL TRIAL: NCT03839290
Title: Three-dimensional Development of the Palate in Bilateral Orofacial Cleft Newborns One Year After Early Neonatal Cheiloplasty: Classic and Geometric Morphometric Evaluation
Brief Title: Development of the Palate in Bilateral Orofacial Cleft Newborns One Year After Early Neonatal Cheiloplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Anthropology and Human Genetics (Unknown); Otorhinolaryngology, 2nd Faculty of Medicine (Unknown); Department of Newborns with Intensive Care Unit (Unknown)
Responsible Party: Principal Investigator, Jana Velemínská, Head of the Department of Anthropology and Human Genetics, Head of Laboratory of 3D Imaging and Analytical Methods, Charles University, Czech Republic
Other Study IDs: 656216
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cleft Palate; Cleft Lip; Cleft Lip and Palate; Cleft Lip, Bilateral
Keywords: bilateral cleft lip and palate; unilateral cleft lip and palate; 3D geometric morphometrics; upper dental arch; classical morphometrics; early neonatal cheiloplasty
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bilateral cleft lip and palate patients: Newborns with complete bilateral cleft lip and palate (cBCLP) and bilateral cleft lip and palate with tissue bridges (BCLP + B) analyzed one year after neonatal cheiloplasty
  Interventions: Procedure: Early neonatal cheiloplasty
- Unilateral cleft lip and palate patients: Newborns with complete unilateral cleft lip and palate (cUCLP) and unilateral cleft lip and palate with tissue bridges (UCLP + B) analyzed one year after neonatal cheiloplasty
  Interventions: Procedure: Early neonatal cheiloplasty

INTERVENTIONS:
Procedure: Early neonatal cheiloplasty

SUMMARY:
Early neonatal cheiloplasty is modified surgery protocol applied in the first week of newborn's life used for treating orofacial cleft patients. This prospective study analyzes the effects of early neonatal cheiloplasty on the growth and development of maxilla and palate during the observed period of one year.

DETAILED DESCRIPTION:
Multidisciplinary treatment of patients with orofacial clefts begins immediately after birth. The first surgical procedure is early neonatal cheiloplasty applied in the first week of the newborn's life, which has been practiced in the Czech Republic for many years. It is a popular parental choice and has a lot of benefits compared to classic cheiloplasty performed between 3-6 months. Unrestricted growth of jaws is essential for the successful therapy of aesthetics and functions. Although there are known a lot of benefits to this surgery, its influence on facial growth is still being studied.

The methodology of this study is based on modern three-dimensional imaging methods and will be evaluated by classic and geometric morphometric analysis of virtual dental models. The existing database includes 137 virtual dental casts (complete and incomplete bilateral or unilateral cleft lip and palate).

The main aim is to verify that the effects of early neonatal cheiloplasty on the facial or palatal growth are minimal in affected individuals and therefore the subsequent development of these structures can be predicted at a later age. Other goals are to evaluate palatal morphology before and one year after early neonatal cheiloplasty, to assess growth of maxilla and palate using classic and geometric morphometry, to assess morphological differences between cleft types and to compare the results with previously published data of neonates operated by later operation protocol and noncleft control groups.

ELIGIBILITY:
Inclusion Criteria:

* Nonsyndromic orofacial cleft
* Czech origin
* Operated by the same surgeon
* Following same surgery protocol (modified Veau surgery protocol)
* Excellent body temperature, blood pressure, oxygen saturation, heart function
* Performing of early neonatal cheiloplasty

Exclusion Criteria:

* Poor health
* Syndromic orofacial cleft
* Operated by later operation protocol (3-6 months)
* Non-Czech origin

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with orofacial clefts operated in the first week of life at the Motol University Hospital in Prague by the same surgeon following the modified Veau surgery protocol.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Growth changes during the first year of life | T0 before early neonatal cheiloplasty (5 ± 5 days) and T1 before palatoplasty (12 ± 6 months).
  Analysis of palatal growth changes in individuals with orofacial clefts after neonatal cheiloplasty (5 ± 5 days) and before palatoplasty (12 ± 6 months).

SECONDARY OUTCOMES:
Comparison of the palatal growth in orofacial cleft patients | 1 year
  Comparison of the growth of the palate in complete and incomplete cleft patients
Differences between cleft types | 1 year
  Morphological differences between complete and incomplete cleft types

CONTACTS AND LOCATIONS:
Overall Officials: Jana Velemínská, Study Director — Department of Anthropology and Human Genetics; Jiří Borský, Study Chair — Department of Otorhinolaryngology; Lenka Jaklová, Study Chair — Department of Anthropology and Human Genetics
Locations (1):
- Lenka Jaklová, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffmannova E, Moslerova V, Dupej J, Borsky J, Bejdova S, Veleminska J. Three-dimensional development of the upper dental arch in unilateral cleft lip and palate patients after early neonatal cheiloplasty. Int J Pediatr Otorhinolaryngol. 2018 Jun;109:1-6. doi: 10.1016/j.ijporl.2018.03.009. Epub 2018 Mar 14. PMID 29728158
- [Background] Hoffmannova E, Bejdova S, Borsky J, Dupej J, Caganova V, Veleminska J. Palatal growth in complete unilateral cleft lip and palate patients following neonatal cheiloplasty: Classic and geometric morphometric assessment. Int J Pediatr Otorhinolaryngol. 2016 Nov;90:71-76. doi: 10.1016/j.ijporl.2016.08.028. Epub 2016 Aug 31. PMID 27729158
- [Background] Jiri B, Jana V, Michal J, Jiri K, Dana H, Miroslav T, Milos C, Zdenek K, Jaroslav F, Jan J, Jiri Z, Renata P, Miroslav P. Successful early neonatal repair of cleft lip within first 8 days of life. Int J Pediatr Otorhinolaryngol. 2012 Nov;76(11):1616-26. doi: 10.1016/j.ijporl.2012.07.031. Epub 2012 Aug 18. PMID 22906307